CLINICAL TRIAL: NCT07331207
Title: The The Effect of 3D Printed Framework Bone-Borne Rapid Maxillary Expander in Young Adults: a CBCT Study
Brief Title: The Effect of 3D Printed Framework Bone-Borne Rapid Maxillary Expander in Young Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohammed Radwan, Dentist Mohammed Radwan, Mansoura University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Mansoura_University
Record Dates: First submitted 2025-12-29; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Bone Anchored Miniscrew Assisted Rapid Palatal Expansion

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- bone anchored miniscrew assisted rapid palatal expansion (Experimental): placement of four mini-screws in the desired location; the 2 anterior mini-implants will be place paramedian in the anterior palate usually around the third Rugae line. The 2 posterior mini-implants will be placed in the alveolar process between the second premolar and first molar roots at approximately 8-9 mm from the gingival margin.
  After that, the device will be retained to the mini-screws by retaining screw.
  Interventions: Device: bone anchored miniscrew assisted rapid palatal expansion

INTERVENTIONS:
Device: bone anchored miniscrew assisted rapid palatal expansion — skeletal rapid maxillary arch expansion

SUMMARY:
Aim of the study: assess the effect of printed framework pure bone-born rapid maxillary expanders on MPS.

Materials and Methods: The intra-oral scan and CBCT will be sent to the lab for MARPE fabrication, four mini-screws size 10mm in length, and 1.7 mm in diameter will be placed, after that, the device will be retained to the mini-screws by retaining screw. The activation of MARPE will be 1 turn (0.25 mm per turn) per day. After 3 months, a CBCT image will be taken to assess the MPS.

Outcomes:

CBCT analysis: For the first premolar and the first molar: points will be made at the most anterior section where the crown and palatal root can be seen at their greatest length. For the second premolar: in the most anterior section showing maximum length of its root. Measuring the distance between the external right and left maxilla edges in the axial view before expansion and after 3 months from the first activation. Tooth inclination will be measured using the coronal section at a point on the most anterior section, where the crown and the mesiobuccal root can be seen at their greatest length. Buccal alveolar bone thickness measurements were made from the outermost point of the bones to the mesiobuccal root at the level of the furcation point, and fenestration were also evaluated.

DETAILED DESCRIPTION:
Aim of the study: to assess the effect of printed framework pure bone-born rapid maxillary expanders on MPS, dental inclination and buccal bone thickness in young adult patients.

Materials and Methods:

Sample size calculation: Sample size calculation was based on effect Effect of 3D Printed Framework Pure Bone-Born Rapid Maxillary Expanders midpalatal suture that was retrived from previous research (Tanga et al. , 2011). Using G power program version 3.1.9.7 to calculate sample size based on effect size of 0,89 using 2-tailed test , α error =0.05 and power = 85%, the total calculated sample size will be 16.

Treatment procedure:

* First visit: Thorough explanation of procedures to the patient, clarifying all details and technical limitations and informing that failure may occur; Taking intra-oral scan (Medit i700).
* The Scan and CBCT will be sent to the lab for MARPE fabrication.
* Second visit: Surgical guide will be placed. After LA infiltration in the palate, a four OrthoEasy Pal mini-screw from Forestadent size 10mm in length, and 1.8 mm in diameter will be placed, using a manual drive attachment for contra-angle handpiece and attached to OrthoEasy blade 10 mm Octagonal.
* After the placement of four OrthoEasy mini-screws in the desired location; the 2 anterior mini-implants will be place paramedian in the anterior palate usually around the third Rugae line, in area commonly described as the T-Zone. The 2 posterior mini-implants will be placed in the alveolar process between the second premolar and first molar roots at approximately 8-9 mm from the gingival margin. as seen in (figure1); device will be placed.
* After that, the OrthoEasy Pal abutments of the device will be retained to the mini-screws by OrthoEasy Pal Retaining screw using blade for OrthoEasy Pal retaining screw for contra-angle handpiece.
* Immediate 2 turns activation will be made in the hyrax after fitting the appliance.
* The activation protocol of MARPE will be 1 turn (0.25 mm per turn) per day.
* The expansion will be completed when the maxillary width overlaps the mandibular width, achieving normal occlusion.
* After 3 months, a CBCT image will be taken to assess the MPS. The rapid maxillary expander will be removed after 3 months period of retention.

Laboratory steps:

1. Scan and CBCT overlapping using OnyxCeph program First the mini screw placed on their position digitally and then fabrication the digital design of MARPE. The process will be completed by printing the design by using (Riton, Dual-150) machine and welding the hyrax to it, followed by finishing and polishing of the device.
2. In the separate step, the surgical guide will be fabricated digitally according to mini screw position

Records:

For all patients the following records are made:

1. Photographs (Extraoral and Intraoral)
2. Upper and lower plaster casts.
3. Radiographs ( Panoramic radiography, Lateral cephalometric and Cone-beam computed tomography systems).

Photographs will be taken 3 times; pre-operative, after MARPE placement and after 3 weeks from the first activation

Cone-beam computed tomography systems (CBCT):

CBCT image (Soredex Cranex 3Dx) will be taken before expansion to record the stage of mid palatal suture and to assess the MPS. Another image will be taken after 3 months from the first activation for evaluating the mid-palatal suture. At the following setting:

- Exposure time: 9 s, 4.0mA, 89kV, field of view [FOV]: 8*15 cm voxel size: 0.32 mm).

According to a previous published research, CBCT scans were taken before expansion (T1) and 1 week after active expansion (T2).

Digital Imaging and Communications in Medicine (DICOM) file image reconstruction and analysis will be performed with OsiriX Lite software.

outcomes:

For CBCT analysis; the following will be determined:

* dimensional reference planes for craniofacial structures orientation and to standardize linear measurements in the axial plane:

  * In the axial plane, the mid-palatine suture will be used.
  * In the mid-sagittal plane. the horizontal palatal plane will be the selected reference
  * In the coronal plane, the image was oriented perpendicular to the patient's midsagittal plane tangent to the most inferior level of nasal floor at the level of first molar where the crown and palatal root can be seen at their greatest length.
* After the image is oriented:

  1. For the pre-expansion images, the axial view will be chosen to determine the maturation stage of MPS and will be recorded.
  2. In both pre-expansion and after 3 months from the first activation images; points will be marked in the axial plane at 3 different locations assisted from coronal plane: first premolar, second premolar and first molar.
* For the first premolar and the first molar: points will be made at the most anterior section where the crown and palatal root can be seen at their greatest length. For the second premolar: in the most anterior section showing maximum length of its root.
* Measuring the distance between the external right and left maxilla edges in the axial view before expansion and after 3 months from the first activation.
* Tooth inclination will be measured using the coronal section (describe for each tooth side R and L) at a point on the most anterior section, where the crown and the mesiobuccal root can be seen at their greatest length. Angle formed by the intersection of two tangents that passes through the central fossa of upper first molar and through the furcation area, to the transversal line at the level of the palate.
* Buccal alveolar bone thickness measurements were made from the outermost point of the bones to the mesiobuccal root at the level of the furcation point

ELIGIBILITY:
Inclusion Criteria:

* Transverse maxillary deficiency with or without crossbite; who requires maxillary expansion
* Age: (18 to 30) years.
* presence of first and second upper premolars and first upper molars
* No previous orthodontic treatment.
* Good oral hygiene and healthy periodontal tissue.
* No significant dentofacial anomalies, any bone defects, or systemic disease.
* Not being pregnant.

Exclusion Criteria:

* previous orthodontic treatment.
* significant dentofacial anomalies, any bone defects, or systemic disease.
* pregnant.
* bad oral hygiene and healthy periodontal tissue.
* loss first and second upper premolars and first upper molars
* growing patients

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2026-06-20 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Tooth inclination | 3 months
  Tooth inclination will be measured using the coronal section (describe for each tooth side R and L) at a point on the most anterior section, where the crown and the mesiobuccal root can be seen at their greatest length. Angle formed by the intersection of two tangents that passes through the central fossa of upper first molar and through the furcation area, to the transversal line at the level of the palate.
mid-palatal suture expansion | 3 months
  Measuring the distance between the external right and left maxilla edges in the axial view before expansion and after 3 months from the first activation.
Buccal alveolar bone thickness | 3 months
  Buccal alveolar bone thickness measurements were made from the outermost point of the bones to the mesiobuccal root at the level of the furcation point

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of dentistry- Mansoura University, Al Mansurah, Egypt